CLINICAL TRIAL: NCT04550442
Title: A Phase I/II Study of Venetoclax in Combination With Azacitidine in Relapsed/Refractory High-Risk Myelodysplastic Syndrome (MDS) or Chronic Myelomonocytic Leukemia (CMML)
Brief Title: Venetoclax and Azacitidine for the Treatment of Relapsed or Refractory High-Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0128; NCI-2020-06538 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0128 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Chronic Myelomonocytic Leukemia; Recurrent Myelodysplastic Syndrome; Refractory Chronic Myelomonocytic Leukemia; Refractory Myelodysplastic Syndrome; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (venetoclax, azacitidine) (Experimental): Patients receive venetoclax PO daily on days 1-14 and azacitidine IV over 15 minutes or SC on days 1-5. Cycles repeat every 4-8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I/II trial investigates the side effects and best dose of venetoclax when given together with azacitidine and to see how well it works in treating patients with high-risk myelodysplastic syndrome or chronic myelomonocytic leukemia that has come back (relapsed) or has not responded to treatment (refractory). Venetoclax may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax and azacitidine together may help to control myelodysplastic syndrome or chronic myelomonocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability (phase 1) and overall response rate (ORR) (phase 2) of venetoclax in combination with azacitidine in patients with high risk myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML) with bone marrow excess blasts > 5% that are relapsed/refractory to prior hypomethylating agent (HMA) therapy.

SECONDARY OBJECTIVES:

I. Rate of complete remission (CR). II. Rate of marrow/morphologic complete remission (mCR). III. Rate of hematologic improvement (HI; erythroid/platelet/neutrophil responses).

IV. Rate of red blood cell (RBC) transfusion independence. V. Rate of platelet (PLT) transfusion independence. VI. Rate of cytogenetic response. VII. Rate of bone marrow blast response. VIII. Time to transformation to acute myeloid leukemia (AML). IX. Duration of response (DOR). X. Overall survival (OS). XI. Progression-free survival (PFS). XII. Time to next MDS treatment (TTNT). XIII. Event-free survival (EFS).

EXPLORATORY OBJECTIVE:

I. To investigate the effects of therapy on MDS and to identify biological markers of response to venetoclax and/or its combination with azacitidine.

OUTLINE: This is a phase I, dose-escalation study of venetoclax followed by a phase II study.

Patients receive venetoclax orally (PO) daily on days 1-14 and azacitidine intravenously (IV) over 15 minutes or subcutaneously (SC) on days 1-5. Cycles repeat every 4-8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days and then every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with post HMA-failure high-risk MDS (Int-2 or high risk by the IPSS with overall score >/=1.5) with excess blasts >5% with failure defined as prior receipt of 4 cycles of HMA therapy with failure to attain a response, or progression of disease or relapse at any time after prior response to HMA therapy.
2. Participants with relapsed/refractory chronic myelomonocytic leukemia (CMML) and therapy-related MDS are also eligible.
3. Hydroxyurea is allowed to lower the white cell count </= 10,000/µl prior to initiation of venetoclax.
4. Adequate hepatic function including total bilirubin ≤ 2.0 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement, and ALT/AST ≤ 3.0 x ULN unless considered due to leukemic involvement.
5. Adequate renal function as calculated using the modified Cockcroft-Gault equation of ≥ 30ml/min, OR creatinine < 2x ULN, unless related to the disease.
6. Signed written informed consent.
7. Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment.
8. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment.
9. Age >/= 18 years of age.
10. ECOG/PS ≤2

Exclusion Criteria:

1. Participants having received any prior BCL2 inhibitor therapy.
2. Participants with MDS with IPSS risk categories Low or Int-1 (overall IPSS score < 1.5).
3. Participants with known HIV infection (due to potential drug-drug interactions between antiretroviral medications and venetoclax). HIV testing will be performed at screening, only if required per local guidelines or institutional standards.
4. Participants known to be positive for hepatitis B or C infection [HCV Ab indicative of a previous or current infection; and/or positive HBs Ag or detected sensitivity on HBV-DNA PCR test for HBc Ab and/or HBs Ab positivity] with the exception of those with an undetectable viral load within 3 months of screening. (Hepatitis B or C testing is not required). Subjects with serologic evidence of prior vaccination to HBV [i.e., HBs Ag-, and anti-HBs+] may participate.
5. Participants has received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of study treatment.
6. Participants has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or Starfruit within 3 days prior to the initiation of study treatment.
7. Participants has a cardiovascular disability status of New York Heart Association Class > 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
8. Participant has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, any other medical condition or known hypersensitivity to any of the study medications including excipients of azacitidine that in the opinion of the investigator would adversely affect his/her participating in this study.
9. Participant has a malabsorption syndrome or other condition that precludes enteral route of administration.
10. Participant exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy (viral, bacterial or fungal).
11. Participant has received a live attenuated vaccine within 4 weeks prior to the first dose of study drug.
12. Participant has a history of other malignancies within 2 years prior to study entry, with the exception of:

    * Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
    * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
    * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent; requires discussion with TA MD.
13. Participant has a white blood cell count > 10 × 109/L. (Hydroxyurea or leukapheresis are permitted to meet this criterion)
14. Female subject has positive results for pregnancy test.
15. Participants with (Grade > 1) unresolved from prior treatment (including chemotherapy, targeted therapy, immunotherapy, experimental agents, radiation, or surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase I) | Up to 28 days
  The MTD is the highest dose level in which < 2 patients of 6 develop first cycle dose-limiting toxicity (DLT).
Overall response rate (ORR) (Phase II) | Up to 5 years post-treatment
  ORR is defined as the proportion of patients who had complete remission (CR), partial remission (PR) or marrow CR (mCR) lasting at least 4 weeks, or hematologic improvement (HI) lasting at least 8 weeks. Will estimate the overall response rate for the combination treatment, along with the 95% credible interval.

SECONDARY OUTCOMES:
Rate of CR | Up to 5 years post-treatment
  The association between CR and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Rate of mCR | Up to 5 years post-treatment
  The association between mCR and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Rate of hematologic improvement | Up to 5 years post-treatment
Rate of platelet transfusion independence | Up to 5 years post-treatment
Rate of red blood cell transfusion independence | Up to 5 years post-treatment
Rate of cytogenetic response | Up to 5 years post-treatment
  The correlation between cytogenetic response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Rate of bone marrow blast response | Up to 5 years post-treatment
  The correlation between bone marrow blast response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Duration of response | The number of days from the date of initial response (PR or better) to the date of first documented disease progression/relapse or death, whichever occurs first, assessed up to 5 years post-treatment
  Will be estimated using the method of Kaplan and Meier. Comparisons by important subgroups will be made using the log-rank tests.
Event-free survival | The number of days from the date of treatment initiation to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first, assessed up to 5 years post-treatment
  Will be estimated using the method of Kaplan and Meier. Comparisons by important subgroups will be made using the log-rank tests.
Overall survival | The time from treatment start till death or last follow-up, assessed up to 5 years post-treatment
  Will be estimated using the method of Kaplan and Meier. Comparisons by important subgroups will be made using the log-rank tests.
Progression free survival | The time from treatment to progression or last follow-up, assessed up to 5 years post-treatment
  Will be estimated using the method of Kaplan and Meier. Comparisons by important subgroups will be made using the log-rank tests.
Time to transformation to acute myeloid leukemia (AML) | The time from treatment till transformation of AML or last follow-up, assessed up to 5 years post-treatment
  Will be estimated using the method of Kaplan and Meier. Comparisons by important subgroups will be made using the log-rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://www.mdanderson.org